CLINICAL TRIAL: NCT04730960
Title: Comparison of Cervical Region Characteristics of People With Smartphone Addiction According to Gender
Brief Title: Comparison of Cervical Region Characteristics of People With Smartphone Addiction
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HATİCE ÇETİN, Research Assisstant, Hacettepe University
Other Study IDs: SP123
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2021-05

CONDITIONS: Neck Pain; Postural; Defect; Young Adult; Technology
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Healthy patients between the ages of 18 and 30 without neck problems will be included in the study.

SUMMARY:
In healthy participantsng adults, the anterior tilt position of the head and consequently flattening of the cervical lordosis may results in impaired neutral posture of the spine during daily long-term computer etc. use with today's technology. In addition, the increasing use of smart phones may also promote this negative results. According to a study, the estimated total smartphone sales for 2012 was 660 million, but as of 2015, it is estimated that a total of one billion units worldwide. It is also thought that phone sales will continue to increase over the years, as it facilitates daily life activities.

As a result of our literature review, the investigators have not come across a study that evaluates demographic information such as the duration of using smartphones or computers, cervical position sense, neck muscle strength, physical activity and general psychological status, which the investigators think may affect the performance of deep cervical flexor muscles in healthy participantsng adults. With this study, it will be ensured that more information about the factors affecting the performance of deep cervical flexor muscles will be determined in advance and necessary steps will be taken to prevent the factors that may cause neck problems in the future.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 18-30,
* Not having mental - cognitive problems,
* Being a volunteer participant.

Exclusion Criteria:

* Having any surgery on the vertebral column,
* Having an inflammatory disease,
* Having a rheumatological disease,
* Having a history of malignancy,
* Having congenital spinal cord anomalies, congenital and / or subsequent spinal deformities,
* Having radiculopathy, myelopathy and / or other neurological disorders, vestibular disorders,
* Having a history of acute trauma.

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Healthy patients between the ages of 18 and 30 without neck problems will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Muscle Strength Assessment | 10-15 minutes
  The strength of the cervical flexor and extensor muscles will be measured with a digital hand dynamometer. While measuring with a dynamometer, the positions and methods of the fine muscle test defined by Lovett will be based on. Each muscle test with the dynamometer will be done three times. The subject will be given a break of at least one minute to rest between repetitions. The highest 3-repetitive results obtained as a result of these measurements will be recorded as the maximum power and in Newton (N) to be used in statistical analysis.
Cervical Joint Range of Movement Assessment | 10-15 minutes
  Cervical Range of Motion (CROM 3) device will be used for active evaluation of cervical range of motion. CROM 3 is a valid and reliable device . The CROM 3 instrument is a special version of the universal goniometer adapted to the cervical region, developed to evaluate cervical joint motion in 3 planes. Flexion and extension range of motion is measured on the first gravity-dependent quadrant on the side of the CROM 3 device. The gravity-dependent second quadrant CROM 3 device is located on the anterior surface and measures the degree of lateral flexion. The third quadrant is a compass dial on the upper surface of the CROM 3 device and measures the right and left rotation. In order for the compass dial to measure the degree of rotation accurately, magnetic field reinforcement, which is a part of the device, was applied to the shoulders of the subject. Flexion, extension, lateral flexion and rotation movements will be measured with the CROM 3 device.
Cervical Joint Position Sense Assessment | 10-15 minutes
  When evaluating joint position sense, 6 positions will be evaluated including flexion, extension, right and left lateral flexion, right and left rotation. CROM 3 device will be used while making measurements. When the subject starts the test, he will be told to sit upright in a comfortable position with the arms at the sides and look forward. The head of the subject will be brought to the targeted point, slowly and passively, up to 65 percent of the maximum range of motion he has, which was previously determined by the physiotherapist. The case will be passively held at the point reached for three seconds and will be told to feel position. Then the head of the subject will be brought back to the neutral position. Then he will be told to remember the phenomenon and passively come to the point brought. The degree of error between the point and the previously determined reference point will be recorded. This process will be repeated three times and the average value will be calculated.
Smartphone Addiction Assessment | 10-15 minutes
  Individuals' smartphone use will be evaluated with the Smartphone Addiction Scale. Kwon et al. The "Smartphone Usage Scale" developed by "Smartphone Usage Scale" is a 6 point Likert type scoring scale consisting of 33 items. Each item is evaluated as "1: Absolutely no" and "6: Absolutely yes". The total score in the scale, which was validated in Turkish, varies between 33-198, and as the score increases, it means increase in smartphone addiction. Daily life disorders consist of 6 subtitles: positive expectation, feeling of deprivation, virtual oriented relationship, overuse and endurance.
Posture Assessment | 10-15 minutes
  Individuals' head and shoulder posture will be evaluated by taking sagittal plan photographs; shoulder and head angles will be calculated. In previous studies, anterior tilt was defined as the angle between the line between the tragus and C7 and the line drawn in the vertical direction from C7 equal to or greater than 46 °. Shoulder protraction is defined as the angle between the line between the acromion and the line C7 and the line drawn vertically from C7 is equal to or greater than 52 °.Reflective markers will be placed on the dominant side ear (tragus), acromion and C7 spinous process; their places will be marked on the skin and in the photo. Individuals will be taught to position them with their feet shoulder-width apart, standing 40 cm in front of the wall, and moving their upper and lower extremities, in their own resting positions. In the sagittal plane, a high resolution digital camera will be placed on a tripod three meters away.
Physical Activity Assessment | 10-15 minutes
  Physical activity levels of individuals will be evaluated with IPAQ - short form. IPAQ - short form consists of 4 separate parts and 7 questions in total. This form contains questions about physical activities performed for at least 10 minutes in the last 7 days. The questionnaire determines how many days in the last week and how long for each day heavy physical activities, moderate intensity physical activities, walking and the time spent during the day without moving (sitting, lying, etc.). It is done by MET method to determine the level of physical activity. The IPAQ - short form has been validated in Turkish.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Cetin, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)